CLINICAL TRIAL: NCT07003152
Title: Prevalence of Endolymphatic Hydrops Among Patients With Hydrocephalus
Brief Title: Relationship Between Hydrocephalus and Endolymphatic Hydrops
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Abdelrahman Abdelghafar, Resident doctor, Sohag University
Other Study IDs: Soh-Med-25-5-5MS
Record Dates: First submitted 2025-05-25; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Hydrocephalus
Keywords: Hydrocephalus, endolymphatic hydrops
MeSH Terms: conditions — Hydrocephalus; Endolymphatic Hydrops

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients with hydrocephalus ages range from 20-60 years including male and female patients: male and female adult patients with hydrocephalus and exclusion criteria were: History of ear diseases, history of Diabetes mellites, or Hypertension, history of Ototoxic drug intake, Congenital anomalies of the auricle or external auditory meatus, history of hereditary hearing loss in the family, noise exposure, other neurological problems apart from hydrocephalus
  Interventions: Diagnostic Test: diagnosis of endolymphatic hydrops in hydrocephalus patients

INTERVENTIONS:
Diagnostic Test: diagnosis of endolymphatic hydrops in hydrocephalus patients — the hydrocephalus could be associated with endolymphatic hydrops, this study designed to show the relationship between both of these diseases by special tests for diagnosis

SUMMARY:
The goal of this observational study is to assess the prevalence of endolymphatic hydrops in patients with hydrocephalus and assess the auditory functions in patients with hydrocephalus including male and female with 20-60 year age groups. it aims to assess the prevalence of endolymphatic hydrops in patients with hydrocephalus and to assess the auditory functions in patients with hydrocephalus

ELIGIBILITY:
Inclusion Criteria: Patients will be diagnosed with hydrocephalus through the neurosurgery department of the same hospital,

Exclusion criteria:

* History of ear diseases
* History of DM or Hypertension
* History of Ototoxic drug intake.
* Congenital anomalies of the auricle or external auditory meatus.
* History of hereditary hearing loss in the family
* History of noise exposure
* Other neurological problems apart from hydrocephalus

Exclusion Criteria:

-

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: hydrocephalic patients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
hearing assessment | 16 weeks
  pure-tone audiometry (air conduction and bone conduction) will be done in a clinical soud-isolatedaudiometry room using two-channel diagnostic audiometer model otopront (90 D-65329 Hohenstein, Germany)